CLINICAL TRIAL: NCT05489913
Title: The Effect of Web Based Cardiac Rehabilitation Support on the Healthy Lifestyle Behaviors, Medication Adherence and Quality of Life in Coronary Artery Patients
Brief Title: Web Based Cardiac Rehabilitation Support in Coronary Artery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semiha ALKAN KAYHAN (Other)
Responsible Party: Sponsor-Investigator, Semiha ALKAN KAYHAN, Nurse, Karadeniz Technical University
Organization: Karadeniz Technical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24237859-534
Record Dates: First submitted 2022-08-01; First posted 2022-08-05 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Cardiac Rehabilitation; Healthy Lifestyle; Medication Adherence; Quality of Life; Coronary Artery Disease
MeSH Terms: conditions — Medication Adherence; Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web based Cardiac Rehabilitation program and follow-up telephone (Experimental): The website was created under the name of "Cardiac Rehabilitation Support Program". The language of the website is Turkish. Designed for computer, tablet and mobile phone use. Patients must be registered to access the website. After creating a six-digit password during registration, they log in to the website with their e-mail address and this password. The password is determined specifically for the patient. There is a welcome text on the home page of the website. The main headings in the menu section; trainings, disease management questions, questionnaires, ask questions to the researcher.
  Interventions: Other: cardiac rehabilitation support program
- Standard care (No Intervention): patients received their training before discharge from the hospital and no intervention was made for 12 weeks.

INTERVENTIONS:
Other: cardiac rehabilitation support program — First of all, a preliminary interview was made with the patients in the experimental group, and their information needs were evaluated individually. Which trainings he should receive and his priorities were determined with the patient. After the training requirements were determined, the general introduction of the website was made and they were allowed to register. Experimental group patients received both training on the website and counseling over the phone for 12 weeks after they started working. A total of 3 phone calls were made with the patients in the first week, 4th and 8th weeks. The interviews lasted an average of 20 minutes. In each phone call, patients were informed and reminded. When patients needed, an average of 2-3 more phone calls were made and information was provided on the subjects they needed.
  Arms: Web based Cardiac Rehabilitation program and follow-up telephone

SUMMARY:
This study was carried out as a randomized controlled experimental study to evaluate the effect of web-based cardiac rehabilitation support on the healthy lifestyle behaviors, medication adherence and quality of life in coronary heart patients.

DETAILED DESCRIPTION:
Hypothesis 1:

H0: Web-based cardiac rehabilitation support has no effect on increasing the healthy lifestyle behaviors of patients with coronary artery disease.

H1: Web-based cardiac rehabilitation support has an effect on increasing the healthy lifestyle behaviors of patients with coronary artery disease.

Hypothesis 2:

H0: Web-based cardiac rehabilitation support in patients with coronary artery disease has no effect on increasing the compliance of patients to drug therapy.

H1: Web-based cardiac rehabilitation support in patients with coronary artery disease has an effect on increasing the compliance of patients to drug therapy.

Hypothesis 3:

H0: Web-based cardiac rehabilitation support has no effect on improving the quality of life of patients with coronary artery disease.

H1: Web-based cardiac rehabilitation support has an effect on improving the quality of life of patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of Coronary artery disease, adult patients, those for whom no surgical operation was planned, those who were clinically stable, those who were literate, those who could communicate verbally, use the Internet, those who had a computer, tablet or smartphone, and those who agreed to participate in the study.

Exclusion Criteria:

* Those who have a disease that is not suitable for the CR program, those who did not agree to participate in the study, those who did not log in after registering on the website, did not read the trainings and could not communicate with the patient during the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Comparison of the total and sub-dimension total scores of the healthy lifestyle behaviors scale of the patients in the experimental and control groups | twelve weeks
  Healthy Lifestyle Behaviors Scale II: The scale has 52 items and six factors.The lowest score obtained from the scale is 52, and the highest score is 208.Healthy lifestyle behaviors score is obtained from the overall score of the scale.High scores obtained from the scale indicate a high level of healthy lifestyle behaviors.
Comparison of experimental and control group patients' compliance with medication adherence | twelve weeks
  Medication Adherence Questions:
  There are three questions in order to evaluate the patients' compliance with drug therapy. These; It consists of questions such as "Do you have problems remembering to take your medicine regularly, do you stop taking your medicine without your doctor's advice when your complaints subside/end, if you don't feel well when you take your medicine (side effects etc.) do you stop taking your medicine?"
Comparison of general quality of life scale index and general quality of life scale vas scores of experimental and control group patients | twelve weeks
  EQ-5D General Quality of Life Scale: It was developed by the Western European Quality of Life Research Society. It consists of five dimensions. In these five dimensions; mobility and walking or walking, doing daily activities with normal daily activities, feeling of pain/discomfort and anxiety/depression and feeling anxious, etc. are evaluated. For the answers given to each dimension, there is no problem, there is some problem, and major problem options are included. A score between -0.59 and 1 is calculated from the five dimensions of the scale. A value of 0 is death, a value of 1 is perfect health, negative values are unconscious and bedridden, etc. points to the results. The scale also includes an easily understandable version of the rated Visual Analog Scale (VAS). Here, participants rate their overall health status from 0 to 100. A score of 100 represents the best health imaginable, while 0 represents the worst.
Comparison of international physical activity questionnaire total scores and physical activity levels of experimental and control group patients | twelve weeks
  International Physical Activity Questionnaire-Short Form: In the scale, walking for at least 10 minutes in the last 7 days, moderate-intensity and intense activities, and sedentary time spent in an average day are asked and metabolic equivalent (MET) scores are calculated. Total time (minutes) and frequency (days) are required to calculate the score. Results are evaluated in three categories: low level, intermediate level and high level. The low level is evaluated as <600 MET, the intermediate level 600-3000 MET, and the high level >3000 MET. The acceptable value in terms of health is expressed as intermediate level, ie 600-3000 MET.
Comparison of body mass index values of experimental and control group patients | twelve weeks
  The formula used to calculate the body mass index is as follows: height (cm)/weight (kg)*weight (kg). After calculating the body mass index of each patient according to this formula, the data were compared.
Comparison of LDL values of experimental and control group patients | twelve weeks
Comparison of smoking status of experimental and control group patients | twelve weeks
  In the patient information form, patients were asked whether they smoked or not.
Post-test Computer System Usability Questionaire Short Version total and sub-dimension scores of the experimental group patients | twelve weeks
  Availability of a computer system; system usefulness (items 1-6), information quality (items 7-9), and interface dimensions (items 10-12) with 13 items. Each item is scored as 1 (strongly agree) and 7 (strongly disagree). The scale was set up in reverse, and low scores indicate good usability of the system.
Comparison of triglyceride values of experimental and control group patients | twelve weeks

CONTACTS AND LOCATIONS:
Overall Officials: Semiha ALKAN KAYHAN, Principal Investigator — ahi Evren thoracic and cardiovascular surgery training and research hospital
Locations (1):
- Health Science University Ahi Evren thoracic and cardiovascular surgery training and research hospital, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No